CLINICAL TRIAL: NCT04325919
Title: Comprehensive Clinical, Virological, Microbiological, Immunological and Laboratory Monitoring of Patients Hospitalized With Coronavirus Disease 2019 (COVID-19)
Brief Title: Coronavirus Disease 2019 (COVID-19) Study of Hospitalized Patients in Hong Kong
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Paul KS Chan, Professor, Chinese University of Hong Kong
Other Study IDs: COVID-19 study 2020.076
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus Infections
Keywords: SARS-CoV-2; Coronavirus disease 2019
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
COVID-19 may cause another world-wide epidemic. This study is divided into 2 arms: (1) Prospective longitudinal observational study involving patients with laboratory-confirmed COVID-19 and (2) Retrospective study on patients with laboratory-confirmed COVID-19.

Arm 1:

We will collect EDTA blood, stool samples, rectal swab, urine, saliva, and specimens from upper respiratory tract (nasopharyngeal aspirate or flocked swab), and lower respiratory tract (sputum or tracheal aspirate) on daily, alternate day, or weekly basis as appropriate.

Arm 2:

The remainder of specimens that were submitted for laboratory investigation as part of clinical management will be retrieved. Those specimens will only be used after all clinically indicated testing and confirmation procedures have been completed. Assistance from the Public Health Laboratory Service, Department of Health, will be invited to retrieve samples as well as participate in this study.

Patients hospitalized for pneumonia in medical wards and ICU at the Prince of Wales Hospital tested negative for COVID-19 will be recruited as controls.

Understanding the clinical, virological, microbiological and immunological profiles of this infection is urgently needed to facilitate its management and control.

ELIGIBILITY:
Inclusion Criteria:

* Case are adults age ≥ 18 years old admitted to hospital with laboratory confirmed COVID-19
* Controls are patients admitted for community-acquired pneumonia

Exclusion Criteria:

* Patients who refuse to consent for study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with laboratory-confirmed COVID-19 in the Prince of Wales Hospital, Princess Margaret Hospital, United Christian Hospital, North District Hospital, Alice Ho Miu Ling Nethersole Hospital, Pamela Youde Nethersole Eastern Hospital, Ruttonjee Hospital, Queen Elizabeth Hospital, and may extend to other hospitals when more cases are detected. The Public Health Laboratory Service, Department of Health, will be invited to assist specimen retrieval and participate in this study.
  Patients hospitalized for pneumonia in medical wards and ICU at the Prince of Wales Hospital tested negative for COVID-19 will be recruited as controls.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-17 (Estimated)

PRIMARY OUTCOMES:
Clinical | 6 months
  Patients' treatment and management during hospitalization.
Virological | 6 months
  Serial viral load changes during hospitalization.
Microbiological | 6 months
  Alterations in fecal microbiota composition (including virome, bacteria and fungi) in COVID-19 patients compared with healthy controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided